CLINICAL TRIAL: NCT00106704
Title: A Multicenter, Randomized, Double Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of the Addition of MK0431 to Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Glimepiride Alone or in Combination With Metformin
Brief Title: Sulfonylurea Add-on Study in Patients With Type 2 Diabetes Mellitus (0431-035)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-035; 2005_009
Record Dates: First submitted 2005-03-29; First posted 2005-03-30 (Estimated); Results first posted 2010-12-17 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Sitagliptin (Experimental): Sitagliptin 10 mg tablet daily for 54 weeks
  Interventions: Drug: Comparator: Sitagliptin
- Placebo/ Pioglitazone (Placebo Comparator): Placebo tablet daily for 24 weeks followed by Pioglitazone tablet daily for 30 weeks
  Interventions: Drug: Comparator: Placebo; Drug: Comparator: Pioglitazone

INTERVENTIONS:
Drug: Comparator: Sitagliptin — sitagliptin 10 mg tablet, once daily for 54 weeks
  Arms: Sitagliptin
Drug: Comparator: Placebo — Placebo oral tablet once daily for 24 weeks
  Arms: Placebo/ Pioglitazone
Drug: Comparator: Pioglitazone — Pioglitazone 30 mg tablet once daily for 30 weeks
  Arms: Placebo/ Pioglitazone

SUMMARY:
The purpose of this clinical study is to determine the safety and efficacy of an investigational drug in patients with Type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 Diabetes Mellitus with inadequate glycemic control

Exclusion Criteria:

* Patients with Type 1 Diabetes Mellitus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2005-03; Primary Completion 2006-06 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Hermansen K, Kipnes M, Luo E, Fanurik D, Khatami H, Stein P; Sitagliptin Study 035 Group. Efficacy and safety of the dipeptidyl peptidase-4 inhibitor, sitagliptin, in patients with type 2 diabetes mellitus inadequately controlled on glimepiride alone or on glimepiride and metformin. Diabetes Obes Metab. 2007 Sep;9(5):733-45. doi: 10.1111/j.1463-1326.2007.00744.x. Epub 2007 Jun 26. PMID 17593236

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 27-Apr-2005. Last Patient Last Visit: 09-Jan-2007. 27 medical clinics in the United States (US), 25 in 11 countries in Europe, and 22 in 11 countries in the rest of the world.
Pre-assignment Details: Patients 18-75 years of age with type 2 diabetes mellitus (T2DM) with inadequate glycemic control (hemoglobin A1c [A1C] ≥7.5% and ≤10.5%) at screening or after treatment with glimepiride (≥4 mg) alone or in combination with metformin (≥1500 mg) for a dose stable period of up to 10 weeks were eligible to participate.
Groups:
- Sitagliptin: The Sitagliptin group includes data from patients randomized to receive treatment with oral tablets of sitagliptin 100 mg q.d. (once daily) with glimepiride (≥4 mg/day) alone or in combination with metformin (≥1500 mg/day).
- Placebo/ Pioglitazone: The Placebo group includes data from patients randomized to receive treatment with placebo to sitagliptin oral tablets q.d. with glimepiride (≥4 mg/day) alone or in combination with metformin (≥1500 mg/day).
Period: Overall Study
Arm/Group | Sitagliptin | Placebo/ Pioglitazone
Started | 222 | 219
Completed | 91 | 68
Not Completed | 131 | 151
Not completed — Adverse Event | 10 | 7
Not completed — Death | 2 | 1
Not completed — Lack of Efficacy | 67 | 69
Not completed — Lost to Follow-up | 7 | 3
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Violation | 4 | 7
Not completed — Withdrawal by Subject | 14 | 21
Not completed — Patient moved | 1 | 0
Not completed — Site terminated | 0 | 1
Not completed — Planned major surgery | 1 | 0
Not completed — Patient Received Glycemic Medication | 22 | 41
Not completed — Unable to re-enter US | 1 | 0
Not completed — Laboratory test | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo/ Pioglitazone | Total
Number analyzed (Participants) | 222 | 219 | 441
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (9.6) | 56.5 (9.6) | 56.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 102 | 207
  Male | 117 | 117 | 234
Race/Ethnicity, Customized [Number; unit: participants]
  White | 136 | 140 | 276
  Black | 10 | 12 | 22
  Hispanic | 39 | 32 | 71
  Asian | 22 | 25 | 47
  Other | 15 | 10 | 25
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 180.9 (37.7) | 181.6 (42.5) | 181.2 (40.1)
Hemoglobin A1C (A1C) [Mean (Standard Deviation); unit: Percent] | 8.34 (0.76) | 8.34 (0.74) | 8.34 (0.75)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at Week 24
Description: Hemoglobin A1C (A1C) is measured as percent. Thus this change from baseline reflects the Week 24 A1C percent minus the Week 0 A1C percent.
Time Frame: Baseline and 24 Weeks
Population: All Patients Treated included patients who received at least 1 dose of study therapy, and had a baseline value and ≥1 post-baseline value for this outcome. The last post-baseline observed measurement was carried forward to Week 24 for patients with no data at Week 24. Data obtained after glycemic rescue were considered missing.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin | Placebo/ Pioglitazone
Number analyzed (Participants) | 217 | 208
Percent | -0.45 [-0.57 to -0.34] | 0.28 [0.17 to 0.40]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo/ Pioglitazone; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, stratum (on metformin or not), baseline A1C; Mean Difference (Net) = -0.74, 95% CI 2-sided [-90.0 to -0.57], Standard Error of Mean 0.08

2. Secondary Outcome: Change From Baseline in FPG at Week 24
Description: The change from baseline is the Week 24 Fasting Plasma Glucose (FPG) minus the Week 0 FPG.
Time Frame: Baseline and 24 Weeks
Population: All Patients Treated included patients who received at least 1 dose of study therapy, and had a baseline value and ≥1 post-baseline value for this outcome. The last post-baseline observed measurement was carried forward to Week 24 for patients with no data at Week 24. Data after rescue were considered missing.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo/ Pioglitazone
Number analyzed (Participants) | 219 | 213
mg/dL | -4.4 [-10.2 to 1.4] | 15.7 [9.8 to 21.6]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo/ Pioglitazone; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, stratum (on metformin or not at Visit 3), baseline A1C; Mean Difference (Net) = -20.1, 95% CI 2-sided [-28.4 to -11.8], Standard Error of Mean 4.2

ADVERSE EVENTS:
Time Frame: Weeks 0 to 54
Description: Patients received glycemic rescue medication if they met specific glycemic goals. SAEs includes events that occurred either before or after receiving rescue medication. Other AEs only includes those AEs that occurred prior to a patient receiving rescue medication.
Arm/Group | Sitagliptin | Placebo/ Pioglitazone
Serious Adverse Events (participants affected / at risk) | 17/222 | 13/219
Other Adverse Events (participants affected / at risk) | 66/222 | 57/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=222) | Placebo/ Pioglitazone (N=219)
Angina Pectoris (Cardiac disorders) | 2 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 2 | 1
Coronary Artery Occlusion (Cardiac disorders) | 1 | 0
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1
Myocardial Ischaemia (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Drowning (General disorders) | 1 | 0
Multi-Organ Failure (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Diabetic Foot Infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Polytraumatism (Injury, poisoning and procedural complications) | 1 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Glioblastoma Multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small Cell Lung Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebellar Infarction (Nervous system disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Completed Suicide (Psychiatric disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=222) | Placebo/ Pioglitazone (N=219)
Nasopharyngitis (Infections and infestations) | 19 | 12
Upper Respiratory Tract Infection (Infections and infestations) | 17 | 20
Urinary Tract Infection (Infections and infestations) | 12 | 6
Blood Glucose Increased (Investigations) | 6 | 11
Hypoglycaemia (Metabolism and nutrition disorders) | 30 | 13
Headache (Nervous system disorders) | 14 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.